CLINICAL TRIAL: NCT01452490
Title: Study of the V-Raser Diode Laser System in the Treatment of Onychomycosis
Brief Title: Diode Laser Treatment of Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConBio, a Cynosure Company (Industry)
Responsible Party: Sponsor
Organization: Cynosure, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: D4-11-F
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Toenail Fungus
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Intervention Model Description: Even though this study has recruited more than 10 participants, it is a feasibility study, designed to test the prototype rather than measuring health outcomes. It is to confirm the operating specifications before beginning a full clinical trial.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diode Laser Treatment (Experimental)
  Interventions: Device: Diode Laser Treatment

INTERVENTIONS:
Device: Diode Laser Treatment — Laser treatment once every 6 weeks, for a total of 4 treatment sessions
  Other Names: V-Raser

SUMMARY:
The purpose of this study is to evaluate the V-Raser diode laser system with investigational Nail Fungus Handpiece in the treatment of onychomycosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed subungual onychomycosis in a great toe that does not extend to the eponychium
* Fitzpatrick Skin Type I-IV
* Written and verbal informed consent
* Able to comply with study instructions and to return to the clinic for required visits
* Agrees to refrain from other active topical, laser or light-based treatment to the great toes
* Agrees to the use of Naftin Gel between the toes to prevent/control tinea pedis

Exclusion Criteria:

* Pregnancy, breastfeeding or planning to become pregnant
* History of cutaneous photosensitivity, porphyria and hypersensitivity to porphyrins or photodermatoses
* Any skin pathology or condition that could interfere with the evaluation or that requires the use of interfering topical or systemic therapy
* Coagulation disorder or current use of anti-coagulation medication (including aspirin use of greater than 81 mg per day)
* Any condition which, in the investigator's opinion, would make it unsafe for the subject to participate
* Enrolled in an investigational drug or device trial, or has been treated with an investigational device or received an investigational drug within 30 days
* Oral Lamisil within 1 year, Sporanox or over-the-counter topicals within 1 month, or other prescription anti-fungal medications or topicals within 6 months
* Evidence of diabetic neuropathy or peripheral vascular disease related to diabetes, or a loss of protective sensation in the affected foot
* Psoriasis, lichen planus, infection involving the lunula, prior surgical treatment of the affected great toe within 1 year, or a history of trauma to the affected great toe
* Immunocompromised status, or with existing (or history of) cancer/skin malignancy
* Distal nail thickness of greater than 2mm in the affected great toenail

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Amount of Clear Nail Growth from Baseline in mm or as measurement of total area of involvement | 12 months
  Amount of lesion-free toenail growth (mm or total area of involvement) from Baseline, as judged by computer software analysis of photos.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Courtright, DPM, Principal Investigator — Shoreline Foot and Ankle Center
Locations (2):
- United States (2):
  - Shoreline Foot and Ankle Center, New London, Connecticut
  - Shoreline Foot and Ankle Center, Westbrook, Connecticut